CLINICAL TRIAL: NCT02667509
Title: The Evolutionary Model of Mild-to-moderate Myopia in China
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Erping Long, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China2
Record Dates: First submitted 2016-01-24; First posted 2016-01-29 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Refractive Error
Keywords: Evolutionary Model
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Myopia has emerged as a major health issue in east Asia, because of its increasingly high prevalence in the past few decades (now 80-90% in school-leavers), and because of the sight-threatening pathologies associated with high myopia, which now aff ects 10-20% of those completing secondary schooling in this part of the world. Similar, but less marked, changes are occurring in other parts of the world. The higher prevalence of myopia in east Asian cities seems to be associated with increasing educational pressures, combined with life-style changes, which have reduced the time children spend outside.

DETAILED DESCRIPTION:
Myopia has emerged as a major health issue in east Asia, because of its increasingly high prevalence in the past few decades (now 80-90% in school-leavers), and because of the sight-threatening pathologies associated with high myopia, which now aff ects 10-20% of those completing secondary schooling in this part of the world. Similar, but less marked, changes are occurring in other parts of the world. The higher prevalence of myopia in east Asian cities seems to be associated with increasing educational pressures, combined with life-style changes, which have reduced the time children spend outside.

In this trial, the investigators aim to study the evolutionary model of myopia in China, which could provide new insight into the social development and human adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Patients complete the examination of Refractive error from 2005 to 2015 year.

Exclusion Criteria:

* Patients could not complete the examination of Refractive error

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects from all the province of China who undergoing the examination of Refractive error from 2005 to 2015 year.
Sampling Method: Probability Sample
Enrollment: 852441 (Actual)
Dates: Start 2005-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Refractive error of both eyes measured by autorefractor and subjective measuring | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin Lin, M.D., Ph.D, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Erping Long, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Morgan IG, Ohno-Matsui K, Saw SM. Myopia. Lancet. 2012 May 5;379(9827):1739-48. doi: 10.1016/S0140-6736(12)60272-4. PMID 22559900
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/